CLINICAL TRIAL: NCT01037842
Title: Phase 3 Study of Combination of Mitiglinide and Metformin in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Combination of Mitiglinide and Metformin on Glycemic Control in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul St. Mary's Hospital (Other); The Catholic University of Korea (Other); Uijeongbu St. Mary Hospital (Other); Korea University (Other); Kyungpook National University Hospital (Other); Pusan National University College of Medicine (Unknown); Sungkyunkwan University (Other); Yonsei University (Other); Eulji University (Other); Chonnam National University (Other); Chonbuk National University (Other); Chungnam National University (Other); Hallym University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMMEDIATE
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mitiglinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin+Mitiglinide (Active Comparator): mitiglinide 10 mg three times a day added to metformin 500 mg three times a day
  Interventions: Drug: Mitiglinide
- Metformin+Placebo (Placebo Comparator): placebo three times a day added to metformin 500 mg three times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mitiglinide — mitiglinide 10 mg three times a day added to metformin 500 mg three times a day
  for 16 weeks
  Arms: Metformin+Mitiglinide
Drug: Placebo — placebo three times a day added to metformin 500 mg three times a day for 16 weeks
  Arms: Metformin+Placebo

SUMMARY:
We performed a prospective, randomized, multicenter trial to assess the efficacy and safety of combined treatment with mitiglinide and metformin for patients with type 2 diabetes who show inadequate glycemic control with metformin monotherapy. Subjects with HbA1c >7.0% after an 8-week metformin run-in phase were randomized to a 16-week trial phase with metformin plus mitiglinide (Met+Mit) or metformin plus placebo (Met).

DETAILED DESCRIPTION:
This was a 16-week, randomized, double-blind study for comparing metformin plus mitiglinide (Met+Mit) versus metformin plus placebo (Met+Pcb). An 8-week metformin run-in phase (500 mg twice a day for the first 4 weeks and 500 mg three times a day for the following 4 weeks) was followed by a 16-week trial phase (mitiglinide 10 mg or placebo three times a day added to metformin 500 mg three times a day). The subjects with an HbA1c >7.0% at the end of the metformin run-in phase were randomized to a Met+Mit group or a Met+Pcb group of the trial phase.

ELIGIBILITY:
Inclusion Criteria:

* aged 30-70 years
* had a duration of diabetes of <10 years
* body mass index (BMI) 20-35 kg/m2
* a plasma HbA1c level of 7.5-11% during the previous 4 weeks

Exclusion Criteria:

* subjects who were diagnosed with type 1 diabetes, gestational diabetes, or diabetes with any specific causes
* Subjects who had been treated with nateglinide, repaglinide, metformin (over 1,000 mg/day), or sulfonylurea (over a quarter of the maximum recommended dose) during the previous 8 weeks

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
the change in HbA1c from randomization to endpoint | 16 weeks after radomization

SECONDARY OUTCOMES:
the proportion of subjects with HbA1c <7% after 16 weeks of treatment and the change in FPG and 2-hr postprandial glucose (PPG) from baseline | 16 weeks after radomization

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Pusan National University College of Medicine, Busan
  - Kyungpook National University School of Medicine, Daegu
  - Chungnam National University College of Medicine, Daejeon
  - Chonnam National University College of Medicine, Gwangju
  - Chonbuk National University College of Medicine, Jeonju
  - Eulji University School of Medicine, Seoul
  - Hallym University College of Medicine, Seoul
  - Korea University College of Medicine, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - SungKyunKwan University School of Medicine, Seoul
  - The Catholic University of Korea, Seoul
  - Yonsei University College of Medicine, Seoul
  - Uijeongbu St. Mary Hospital, Uijeongbu-si